CLINICAL TRIAL: NCT01906541
Title: A Phase I/II Gene Therapy Trial for X-CGD With a SIN Gammaretroviral Vector
Brief Title: Gene Therapy for X-CGD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hubert Serve, Prof., MD (Other)
Responsible Party: Sponsor-Investigator, Hubert Serve, Prof., MD, Head of Medical Department II, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X-CGD
Record Dates: First submitted 2013-07-15; First posted 2013-07-24 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: X-linked Chronic Granulomatous Disease
Keywords: X-CGD; chronic granulomatous disease; gene-therapy
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ex-vivo gene-therapy (Experimental): transplantation of genetically modified autologous CD34+ cells
  Interventions: Genetic: ex-vivo gene-therapy

INTERVENTIONS:
Genetic: ex-vivo gene-therapy — transplantation autologous CD34+ cells, transduced with a SIN gammaretroviral vector

SUMMARY:
X-linked chronic granulomatous disease (X-CGD) is a rare inherited immune defect, which is caused by the inability of phagocytic cells to produce reactive oxygen species due to a defect in the gp91phox subunit of the NADPH oxidase complex. X-CGD patients suffer from recurrent and life-threatening infections and severe hyperinflammatory complications.

The only curative treatment for X-CGD is allogenic hematopoietic stem cell transplantation, but this procedure implies severe risks and many patients lack an appropriate donor. Therefore alternative curative approaches are urgently needed. In this study, patients will be treated with gene-corrected autologous CD34+ cells, using a SIN gammaretroviral vector for ex-vivo gene-therapy.

ELIGIBILITY:
Inclusion Criteria:

* Verified diagnosis of the X-linked form of chronic granulomatous disease, with loss of gp91phox expression (Western Blot). Evidence of less than 5% of normal oxidase production in circulating neutrophil granulocytes as measured by dihydrorhodamine- (DHR-) and nitro blue tetrazolium- (NBT-) assay
* History of severe chronic infections with life-threatening course or severe steroid- sensitive or steroid insensitive granulomatous disease, with necessity of inpatient treatment, without sustained improvement even under maximum conservative treatment measures
* No Human Leukocyte Antigen (HLA) identical (10/10 match) sibling- or unrelated donor, or contraindications for allogenic stem cell transplantation in presence of a suitable donor. The lack of an HLA-identical (10/10 match) sibling- or unrelated donor has to be confirmed by an unsuccessful search in national and international donor registers for at leat 3 months
* Normal organ-function: glomerular filtration rate (GFR) ≥ 60ml/min., Bilirubin ≤ 1.5-fold upper reference-level, normal parameters for liver enzymes and clotting (TPZ 75-100%, partial thromboplastin time (PTT) 30-38sec, Fibrinogen 200-400mg/dl), Leukocytes > 3 x 10^9/l, Granulocytes > 1.5 x 10^9/l, Thrombocytes >100 x 10^9/l
* Contraception from start of G-CSF application until 1 year after retransfusion of the gene-corrected cells
* No interferon-gamma injection within two weeks prior to hematopoietic stem cell mobilization
* Karnofsky-Index > 70%
* Signed informed consent

Exclusion Criteria:

* Patients with non-controlled acute infections
* Severe cardiac or pulmonary malfunctions: ejection fraction < 60%, valvular heart disease > II°, arrhythmia requiring therapy, forced expiratory volume at one second/vital capacity (FEV1/VC) < 75% , diffusion capacity of lung for carbon monoxide (DLCO) <60%
* Bilirubin > 1.5-fold upper reference-level
* HIV-, Hepatitis B- or C - infection
* Contraindications for G-CSF administration, as autoimmune vasculitis.
* Contraindications for stem cell apheresis, as low hemoglobin < 8g/dl, cardiovascular instability or severe coagulopathy
* Pregnancy or breast-feeding
* Drug- or alcohol-abuse
* Lack of search for an unrelated donor
* Patients with a HLA 9/10 mismatched unrelated donor (MMUD) will be excluded, if a thorough risk-benefit analysis favors allogenic hematopoietic stem cell transplantation (HSCT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Transduction rate of granulocyte colony-stimulating factor (G-CSF) mobilized peripheral CD34+ cells from CGD patients with a SIN gamma retroviral vector | 1 week
Engraftment rate of the transduced CD34+ cells in the patients | 5 years
Long-term expression of the transgene (rate of gp91phox positive cells) in circulating cells in the peripheral blood | 5 years
Functional reconstitution of the NADPH oxidase in circulating cells of the peripheral blood (% DHR positive cells) | 5 years
Frequency and severity of unexpected toxic adverse events during and after infusion of the genetically modified CD34+ cells | 5 years

SECONDARY OUTCOMES:
Frequency of infections as indicator for the clinical benefit for the patients | 5 years
Proliferation rate of CD34+ cells in ex-vivo culture under serum-free conditions | up to 3 weeks
Differentiation rate of CD34+ cells (as measured by flow cytometry) in ex-vivo culture under serum-free conditions | up to 3 weeks
Transduction rate of CD34+ cells in ex-vivo culture under serum-free conditions | up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Germany